CLINICAL TRIAL: NCT03298737
Title: Visual Attention and Eye Movements
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jude Mitchell, Assistant Professor, University of Rochester
Other Study IDs: RSRB00068408
Record Dates: First submitted 2017-09-20; First posted 2017-10-02 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Vision, Ocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Correct to normal vision population
  Interventions: Behavioral: Covert Spatial Attention

INTERVENTIONS:
Behavioral: Covert Spatial Attention — During behavioral sessions, subjects will sit in a dark room and view a video monitor placed at the minimum of 57 cm distance away from the subject. Staff will be present throughout all the testing to assist the subject and monitor equipment that is used for tracking their eye position. Subjects will be asked to maintain their heads in a stable position of rest in order to insure accurate tracking of their eye position. To stabilize their head, subjects will either use a "chin rest" in which they position their chin on a soft pad mounted in front of a video screen, or they may use a "bite bar."

SUMMARY:
The purpose of this study is to provide information about how the brain processes sensory inputs using visual stimuli throughout various psychophysical experiments.

DETAILED DESCRIPTION:
This laboratory studies visual perception with a focus on the interaction between eye movements and attention. It is well established that attending to a stimulus can profoundly alter perception. For example, attending to a speaker at a crowded party can almost completely filter background both in terms of auditory noise and visual distractions. Although laboratory studies have traditionally investigated the effects of attentional changes in the absence of eye movements, under natural conditions, visual attention is often accompanied by orienting movements to direct our head and eyes towards the relevant objects of interest. Recent work has suggested that these orienting movements affect perception in a manner similar to covert attention. The proposed studies will investigate how eye movements contribute to perception and attention.

The research covered by this protocol combines traditional "button-press" psychophysics with non-invasive eye-tracking to investigate the interaction between eye movements and perception. Subjects will perform simple perceptual tasks, such as judging the orientation or direction of a visual stimulus, while their eye position is monitored with a video eye-tracker. This approach (combining psychophysics and eye-tracking) is flexible, low risk, and fast when compared with neurophysiological studies. However, by focusing on low-level perceptual tasks, the results will be interpretable in the context of larger studies of neurophysiological responses in the visual system.

The investigators hope that this basic research will ultimately have both applied and clinical significance. For example, understanding how perception is influenced by attention and eye-movements in neurotypical populations may provide non-invasive and naturalistic ways to identify and diagnose psychiatric disorders. Additionally, understanding how eye-movements interact with sensory encoding has the potential to improve machine learning algorithms for vision and navigation (These are not a part of the current study, but a potential future impact).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65
* Corrected-to-normal vision
* No known diagnosis of visual or auditory disorder or impairment

Exclusion Criteria:

* Does not have corrected-to-normal vision
* Unable to understand and follow the instructions given of the study
* Known diagnosis of visual or auditory disorder or impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants age 18-65 with corrected to normal vision
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-10-26 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Pursuit eye movements to peripheral moving stimuli | baseline
  Pursuit eye movements are smooth eye movements with slow velocities (< 15 degs/sec) that track the motion of visual stimuli when they are at the center of the visual field (Madelain and Krauzlis, J. of Vision, 2003). Here we will test the prediction that pursuit eye movements begin to track the motion of the stimulus located peripherally as an eye movement moves to the stimulus. The null hypothesis is that there will be no effect of the peripheral stimulus motion on the pursuit eye movements. We will measure eye movements using an infra-red eye tracker (Arrington, Inc) from 500 or more trials collected in each session. The distribution of pursuit eye movements will be computed for each subject to evaluate if there is significant pursuit along the direction of stimulus motion around the time of the saccade. The mean per participant will be determined and group effects evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Brain and Cognitive Sciences, University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madelain L, Krauzlis RJ. Pursuit of the ineffable: perceptual and motor reversals during the tracking of apparent motion. J Vis. 2003 Nov 18;3(11):642-53. doi: 10.1167/3.11.1. PMID 14765950